CLINICAL TRIAL: NCT05797844
Title: Improving the Endotracheal Tube Cuff Pressure Control Management Knowledge of Intensive Care Nurses: A Quasi-Experimental Study Pre-Post Test
Brief Title: Improving the Endotracheal Tube Cuff Pressure Control Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Selda Karaveli Çakır, Assistant professor, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-KAEK-143-59
Record Dates: First submitted 2023-03-03; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Nurse's Role
Keywords: cuff pressure management; endotracheal tube cuff; educational intervention; intensive care nurses; nurses' knowledge
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Nurses included in experimental group were trained through a 4-hour presentation (passive implementation strategy) prepared in the presence of evidence-based guidelines and literature, in addition, they were given a brochure about cuff pressure measurement and a brochure about cuff pressure was hung in the intensive care units where there are handwashing sinks. In addition, 4 follow-up visits (active strategy) were carried out for ETT cuff pressure management using the one-on-one demonstration technique every 21 days.
  Interventions: Other: Active implementational educational strategy; Other: Passive implementational educational strategy
- Control Group (Active Comparator): Nurses included in control group were trained through a 4-hour presentation (passive implementation strategy) prepared in the presence of evidence-based guidelines and literature, in addition, they were given a brochure about cuff pressure measurement and a brochure about cuff pressure was hung in the intensive care units where there are handwashing sinks.No follow-up visits were made to this group
  Interventions: Other: Passive implementational educational strategy

INTERVENTIONS:
Other: Active implementational educational strategy — 4 follow-up visits (active implemantation strategy) were carried out for ETT cuff pressure management using the one-on-one demonstration technique every 21 days. These follow-ups included adherence to evidence-based guidelines, nurses' application of endotracheal cuff pressure measurement and solving the problems encountered during its implementation. Uncertainties associated with evidence-based guidance on endotracheal tube cuff pressure control were clarified during these sessions.
  Other Names: Experimental group
  Arms: Experimental Group
Other: Passive implementational educational strategy — Theoretical training on endotracheal tube cuff pressure management through a 4-hour presentation prepared with evidence-based guide and literature. A PowerPoint presentation including endotracheal tube cuff pressure normal values, complications related to endotracheal tube cuff pressure, management of endotracheal tube cuff pressure, endotracheal tube cuff pressure control methods, methods affecting endotracheal tube cuff pressure, how to measure endotracheal tube cuff pressure was made.
  Other Names: Control group

SUMMARY:
This study aimed to evaluate how an educational intervention based on the existing evidence-based guidelines, using both active and passive educational implementetion strategies, could improve the knowledge of nurses regarding managing ETT cuff pressure control.

Hypothesis H1: There is a difference between the training given with the active and passive implementation strategies method in improving the endotracheal cuff pressure control knowledge of intensive care nurses.

DETAILED DESCRIPTION:
This study was carried out as a quasi-experimental two-group pretest-posttest research design to evaluate the effect of endotracheal tube cuff pressure control training given with the active and passive implementation strategies methods on the knowledge level of nurses. The research was carried out in the intensive care units of a Training and Research Hospital, between June and December 2022, in 6 intensive care units (General ICU 1-General ICU 2- General ICU 3, CVC ICU, 2nd Level ICU, Coronary ICU).

In the intensive care unit of the hospital where the study was conducted, the endotracheal tube cuff pressure is controlled by the pilot balloon finger palpation method in four hours. In addition, pressure measurement was not made with the cuff manometer. However, in endotracheal tube cuff control, cuff pressure should be monitored to prevent aspiration and the cuff pressure should be kept between 20-30 cmH2O. Before the data of the study started to be collected, a cuff manometer was purchased by the hospital management to be used in the intensive care units.

The universe of the research consisted of 120 nurses working in the intensive care units where the study was conducted. The necessary sample of the study was determined by using G*Power computer software program version 3.0.1 as recommended to be used in calculating the desired sample by previous studies. The sample consisted of 90 nurses scheduled for, with a power value to represent 95% of the study population at a 80% confidence interval, 0.05 error level, and 0.6 effect size according to power analysis. Research Randomizer software (http://www.randomizer.org.) was used to generate a randomized list by applying a simple randomization technique to each participant's allocation. The 90 participants were divided into two even groups (Intervention Group =45, Control Group =43 nurses).

Sociodemographic and occupational characteristics form and knowledge level evaluation form regarding endotracheal tube cuff pressure control were used to collect the data of the study.

Since the nurses working in the intensive care unit work in day and night shifts, the sociodemographic and occupational characteristics form to be applied before the training and the knowledge level evaluation form on endotracheal tube cuff pressure control (pretest) were collected by the researchers after the nurses' shift delivery hours. After applying the pre-test questionnaires (experimental /Control group), on the days determined together with the intensive care unit nurses in charge and the nursing services directorate, all nurses were given theoretical training on endotracheal tube cuff pressure management through a 4-hour presentation prepared with evidence-based guide and literature. Thus, all nurses gained equal knowledge. A PowerPoint presentation including endotracheal tube cuff pressure normal values, complications related to endotracheal tube cuff pressure, management of endotracheal tube cuff pressure, endotracheal tube cuff pressure control methods, methods affecting endotracheal tube cuff pressure, how to measure endotracheal tube cuff pressure was made.

Nurses included in experimental group were trained through a 4-hour presentation (passive implementation strategy) prepared in the presence of evidence-based guidelines and literature, in addition, they were given a brochure about cuff pressure measurement and a brochure about cuff pressure was hung in the intensive care units where there are handwashing sinks. In addition, 4 follow-up visits (active implementation strategy) were carried out for ETT cuff pressure management using the one-on-one demonstration technique every 21 days. These follow-ups included adherence to evidence-based guidelines, nurses' application of endotracheal cuff pressure measurement and solving the problems encountered during its implementation. Uncertainties associated with evidence-based guidance on endotracheal tube cuff pressure control were clarified during these sessions. Nurses included in control group were trained through a 4-hour presentation (passive implamentation strategy) prepared in the presence of evidence-based guidelines and literature, in addition, they were given a brochure about cuff pressure measurement and a brochure about cuff pressure was hung in the intensive care units where there are handwashing sinks. No follow-up visits were made to this group. 3 months after the training, the Knowledge Level Evaluation Form (post-test) on Endotracheal Tube Cuff Pressure Control was re-applied to all nurses working in intensive care units and participating in the study.

The results of the study were analyzed in the IBM SPSS Statistics 23.0 (Statistical Package for Social Sciences IBM Corp., Armonk, NYC, USA) package program. Number, percentages, means, standard deviations, were used for descriptive statistics of demographic and occupational characteristics of the nurses. Correct answers to the questions on the knowledge level form were given one point each while incorrect ones were given zero points. The knowledge level scores were calculated by averaging the number of correct answers. The Shapiro-Wilk test was used for normality. The t-test was used to evaluate the education level between the intervention groups before and after the training. The Paired Sample t Test was used to compare the pre-training and post-training average scores for each groups. In all results, p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse in intensive care units
* Nurses who participated in the theoretical training and visited for follow-up
* Volunteer to participate in the study

Exclusion Criteria:

* Not willing to participate in the study
* Forms with missing answers were not included in the evaluation

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
The Knowledge Level Evaluation Form- Pre- test | before theoretical training
  Knowledge level evaluation form on endotracheal tube cuff pressure control consists of 20 questions about the safe limits of endotracheal tube cuff pressure, complications of endotracheal tube cuff pressure that is not within safe limits, the factors affecting endotracheal cuff pressure, and the level of knowledge about endotracheal tube cuff pressure control methods and was prepared by researchers in line with the literature. While creating the survey, expert opinion was obtained. The 20-item knowledge level form was developed to assess the knowledge of nurses on ETT cuff pressure control by researchers. Only one item (part 1) had four answers options the range of ETT cuff pressure, "10-20cmH2O", "20-30 cmH2O", "30-40 cmH2O" and "above 40cmH2 O". Another items had two answers options, "correct" and "incorrect". While scoring, correct answers scored one point each, when incorrect answers options scored zero
The Knowledge Level Evaluation Form-Post-test | 3 months after theoretical training
  Knowledge level evaluation form on endotracheal tube cuff pressure control consists of 20 questions about the safe limits of endotracheal tube cuff pressure, complications of endotracheal tube cuff pressure that is not within safe limits, the factors affecting endotracheal cuff pressure, and the level of knowledge about endotracheal tube cuff pressure control methods and was prepared by researchers in line with the literature. While creating the survey, expert opinion was obtained. The 20-item knowledge level form was developed to assess the knowledge of nurses on ETT cuff pressure control by researchers. Only one item (part 1) had four answers options the range of ETT cuff pressure, "10-20cmH2O", "20-30 cmH2O", "30-40 cmH2O" and "above 40cmH2 O". Another items had two answers options, "correct" and "incorrect". While scoring, correct answers scored one point each, when incorrect answers options scored zero

CONTACTS AND LOCATIONS:
Overall Officials: Selda Karaveli Cakir, Principal Investigator — Kastamonu Universty
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mpasa F, van Rooyen DRM, Venter D, Jordan P, Ten Ham-Baloyi W. Improving nurses' knowledge of managing endotracheal tube cuff pressure in intensive care units: A quasi-experimental study. Health SA. 2020 Dec 18;25:1479. doi: 10.4102/hsag.v25i0.1479. eCollection 2020. PMID 33391829
- [Result] Soyer Ö, Özyürek P, Yavuz van Giersbergen M. The Effect of Endotracheal Tube Cuff Pressure Control Training on Nurses' Knowledge Level. Turk J Intensive Care 2020;18:146-54.
- [Result] Murugiah UR, Ramoo V, Jamaluddin MFH, Yahya A, Baharudin AA, Abu H, Thinagaran RRR. Knowledge acquisition and retention among nurses after an educational intervention on endotracheal cuff pressure. Nurs Crit Care. 2021 Sep;26(5):363-371. doi: 10.1111/nicc.12600. Epub 2021 Feb 10. PMID 33569880